CLINICAL TRIAL: NCT01869725
Title: Comparator Study of 68Ga-DOTATOC PET/CT With Octreoscan + High-resolution, Contrast-enhanced CT for Diagnosis and Staging in Neuroendocrine Tumors and Other Somatostatin Receptor Positive Tumors
Brief Title: Comparative Study of Sensitivity of Ga-DOTATOC PET vs Octreoscan SPECT + CT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sue O'Dorisio (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Sue O'Dorisio, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201212736; NCI-2013-00936 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA086862 (NIH); R01CA167632 (NIH)
Record Dates: First submitted 2013-05-31; First posted 2013-06-05 (Estimated); Results first posted 2021-09-22 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2018-12

CONDITIONS: Adult Medulloblastoma; Childhood Medulloblastoma; Neuroblastoma; Neuroendocrine Tumor; Somatostatinoma
Keywords: Neuroendocrine Tumor; Ga-DOTATOC PET; Imaging
MeSH Terms: conditions — Medulloblastoma; Neuroblastoma; Neuroendocrine Tumors; Somatostatinoma | interventions — gallium Ga 68 dotatate; Magnetic Resonance Spectroscopy; pentetreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (gallium Ga 68-edotreotide PET/CT) (Experimental): Patients receive gallium Ga 68-edotreotide IV and undergo PET/CT scan. Within 120 days, patients undergo standard indium In 111 pentetreotide contrast-enhanced CT or MRI scan. Patients may undergo a second gallium Ga 68-edotreotide PET/CT scan within 3-6 months if the lesions of the first scan cannot be confirmed.
  Interventions: Drug: gallium Ga 68-edotreotide; Procedure: positron emission tomography/computed tomography; Radiation: indium In 111 pentetreotide; Procedure: computed tomography; Procedure: contrast-enhanced magnetic resonance imaging

INTERVENTIONS:
Drug: gallium Ga 68-edotreotide — Given IV
  Other Names: Ga-68 DOTA0-Tyr3-octreotide; Ga-68 DOTATOC
Procedure: positron emission tomography/computed tomography — Undergo gallium Ga 68-edotreotide PET/CT scan
Radiation: indium In 111 pentetreotide — Undergo indium In 111 pentetreotide contrast-enhanced CT or MRI scan
  Other Names: Indium-111 Octreotide DTPA; Indium-111-DTPA-D-Phe-1-octreotide; Indium-In 111 Pentetreotide; Indium-In-111-Pentetreotide; Octreoscan
Procedure: computed tomography — Undergo indium In 111 pentetreotide contrast-enhanced CT scan
  Other Names: tomography, computed
Procedure: contrast-enhanced magnetic resonance imaging — Undergo indium In 111 pentetreotide contrast-enhanced CT or MRI scan
  Other Names: Contrast-enhanced MRI

SUMMARY:
This clinical trial studies gallium Ga 68-edotreotide positron emission tomography (PET)/computed tomography (CT) compared with indium In 111 pentetreotide plus contrast-enhanced CT (or MRI) in diagnosing patients with neuroendocrine tumors and other somatostatin receptor positive tumors. Diagnostic procedures, such as gallium Ga 68-edotreotide PET/CT, may help find and diagnose somatostatin receptor positive neuroendocrine tumors. It is not yet known whether Ga 68-edotreotide PET/CT is as effective as indium In 111 pentetreotide plus contrast-enhanced CT (or MRI) in diagnosis and staging of patients with neuroendocrine tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare efficacy of [68Ga]-DOTA-tyr3-Octreotide (68Ga-DOTATOC) (gallium Ga 68-edotreotide) PET/CT with Octreoscan (indium In 111 pentetreotide) + high-resolution, contrast-enhanced CT for diagnosis and staging in patients with somatostatin receptor expressing tumors.

OUTLINE:

Patients receive gallium Ga 68-edotreotide intravenously (IV) and undergo PET/CT scan. Within 120 days, patients undergo standard indium In 111 pentetreotide contrast-enhanced CT or MRI scan. Patients may also undergo a second gallium Ga 68-edotreotide PET/CT scan within 3-6 months if the lesions of the first scan cannot be confirmed.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Biopsy proven neuroendocrine tumor, neuroblastoma, medulloblastoma, or other somatostatin receptor positive tumor
* Off Sandostatin (octreotide acetate)-long acting release (LAR) > 4 weeks and off immediate release (subcutaneous) for 12 hrs prior to 68Ga-DOTATOC PET-CT
* Karnofsky performance status or Lansky Play Scale status of >= 50 (or Eastern Cooperative Oncology Group [ECOG]/World Health Organization [WHO] equivalent)
* Subject is male; or is a female who is either pre-menarchal, surgically sterile (has had a documented bilateral oophorectomy and/or documented hysterectomy), postmenopausal (> 1 years without menses), non-lactating, or of childbearing potential for whom a serum pregnancy test (with the results known prior to investigational product administration) is negative; a negative serum pregnancy test will be required for all female subjects with child bearing potential; if a false pregnancy test is suspected, e.g., perimenopausal condition, an obstetrician will be consulted to determine if she is/is capable of becoming pregnant
* No therapy other than Sandostatin since last Octreoscan + diagnostic CT
* Fresh frozen (recommended) or paraffin fixed (required) specimen of primary or metastases available for ribonucleic acid (RNA) and immunohistochemistry (IHC)

Exclusion Criteria:

* Pregnancy or breast feeding
* Surgical resection, chemotherapy, radiation therapy, or biologic therapy since last Octreoscan + CT; continuation of the same dose of Sandostatin-LAR or subcutaneous Sandostatin is allowed
* Medical condition uncontrolled by treatment making completion of study unlikely
* Weight more than 400 pounds (subjects who weigh more than 400 pounds will not be able to fit inside the imaging machines)
* Inability to lie still for the entire imaging time (e.g. cough, severe arthritis, etc.)
* Inability to complete the needed investigational and standard-of-care imaging examinations due to other reasons (severe claustrophobia, radiation phobia, etc.)
* Any additional medical condition, serious intercurrent illness, or other extenuating circumstance that, in the opinion of the investigator, may significantly interfere with study compliance

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2018-12-26 (Actual); Study Completion 2018-12-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. Sue O' Dorisio, MD, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diagnostic (Gallium Ga 68-edotreotide PET/CT)
Started | 68
Completed | 64
Not Completed | 4
Not completed — ineligible after registration | 1
Not completed — Death | 1
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: 68 patients enrolled
Arm/Group | Diagnostic (Gallium Ga 68-edotreotide PET/CT)
Number analyzed (Participants) | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5
  Between 18 and 65 years | 45
  >=65 years | 18
Age, Continuous [Mean (Full Range); unit: years] | 55 [4 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 28
  More than one race | 1
  Unknown or Not Reported | 38
Region of Enrollment [Number; unit: eligible participants]
  United States | 68

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Conventional Imaging and Gallium Ga 68-edotreotide PET Using Concordance in Tumor Detection With Pathology
Description: Tumor lesions detected on 68Ga-DOTATOC PET/CT compared with tumor lesions detected on Octreoscan SPECT imaging plus high-resolution, contrast-enhanced CT.
Time Frame: Up to 6 months between the timing of the Octreoscan SPECT/CT plus high-resolution, contrast-enhanced CT and the time of the 68Ga-DOTATOC PET/CT (either imaging type may occur first)
Population: Patients with neuroendocrine tumor or other somatostatin receptor positive tumor
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic (Gallium Ga 68-edotreotide PET/CT)
Number analyzed (Participants) | 34
Participants
  Sensitivity and Specificity for Ga-68-DOTATOC as Compared to Pathology: Total positive | 28
  Sensitivity and Specificity for Ga-68-DOTATOC as Compared to Pathology: False position | 0
  Sensitivity and Specificity for Ga-68-DOTATOC as Compared to Pathology: False negative | 1
  Sensitivity and Specificity for Ga-68-DOTATOC as Compared to Pathology: Total negative | 5
  Sensitivity and Specificity for OctreoScan as Compared to Pathology: Total positive | 23
  Sensitivity and Specificity for OctreoScan as Compared to Pathology: False position | 0
  Sensitivity and Specificity for OctreoScan as Compared to Pathology: False negative | 6
  Sensitivity and Specificity for OctreoScan as Compared to Pathology: Total negative | 5

2. Primary Outcome: Compare Sensitivity of 68Ga-DOTATOC PET/CT With Octreoscan
Description: Compare sensitivity of 68Ga-DOTATOC PET/CT with Octreoscan + high-resolution, contrast-enhanced CT for diagnosis and staging in neuroendocrine tumors and other somatostatin receptor positive tumors
Time Frame: Up to 6 months
Population: Patients with neuroendocrine tumor or other somatostatin receptor positive tumor
Measure: Number; unit: percentage of sensitivity
Arm/Group | Diagnostic (Gallium Ga 68-edotreotide PET/CT)
Number analyzed (Participants) | 34
percentage of sensitivity
  Sensitivity of Ga-68-DOTATOC | 96.55
  Sensitivity of OctreoScan | 79.31
  Sensitivity of Conventional Imaging (CI) | 82.24

3. Primary Outcome: Compare Specificity of 68Ga-DOTATOC PET/CT With Octreoscan
Description: Compare specificity of 68Ga-DOTATOC PET/CT with Octreoscan + high-resolution, contrast-enhanced CT for diagnosis and staging in neuroendocrine tumors and other somatostatin receptor positive tumors
Time Frame: 6 months
Population: Patients with neuroendocrine tumor or other somatostatin receptor positive tumor
Measure: Number; unit: percentage of specificity
Arm/Group | Diagnostic (Gallium Ga 68-edotreotide PET/CT)
Number analyzed (Participants) | 34
percentage of specificity
  Specificity of 68Ga-DOTATOC | 100
  Specificity of Octreoscan | 100
  Specificity of Conventional Imaging (CI) | 47.82

ADVERSE EVENTS:
Time Frame: Adverse events were collected over 6 months at the following time points: 1) screening visit which occurred within 30 days of Ga-68 DOTATOC PET/CT 2) at scan 1 3) 1-7 days post scan 1 4) at scan 2 5) 1-7 days post scan 2
Arm/Group | Diagnostic (Gallium Ga 68-edotreotide PET/CT)
All-Cause Mortality (participants affected / at risk) | 1/68
Serious Adverse Events (participants affected / at risk) | 0/68
Other Adverse Events (participants affected / at risk) | 11/68
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diagnostic (Gallium Ga 68-edotreotide PET/CT) (N=68)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) — cramping
Nausea (Gastrointestinal disorders) | 4 (4)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) — chills
Pain (General disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) — joint stiffness
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Flushing (Vascular disorders) | 2 (2)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1) — skin mottling

LIMITATIONS AND CAVEATS:
Although 67/68 were eligible and received the 68Ga-DOTATOC PET scan, four patients did not receive the 111In-Octreotide SPECT scan. Of the 63 subjects who received both scans, 30 subjects did not receive the 111In-Octreotide SPECT scan within either the six months prior to or six months after the 68Ga-DOTATOC PET scan. This left only 34 subjects who could be fully evaluated for comparison of number of lesions found on both scans.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-03-26): https://cdn.clinicaltrials.gov/large-docs/25/NCT01869725/Prot_SAP_000.pdf
  • Informed Consent Form (2015-02-20): https://cdn.clinicaltrials.gov/large-docs/25/NCT01869725/ICF_001.pdf